CLINICAL TRIAL: NCT00931593
Title: Transient Lower Esophageal Sphincter Relaxations Detection Using High Resolution Manometry. Validation in Healthy Volunteers.
Brief Title: Transient Lower Esophageal Sphincter Relaxations and High Resolution Manometry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Dr Sabine ROMAN, Hospices Civils de Lyon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008.546/47
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-07

CONDITIONS: Healthy Volunteers
Keywords: Transient lower esophageal sphincter relaxation; high resolution manometry; dentsleeve probe; healthy volunteers
MeSH Terms: interventions — Manometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- volunteers (Experimental): This is a descriptive study to compare two techniques (manometry with perfused dentsleeve probe vs high resolution manometry for the identification of tLESr). Each subject is his own control.
  The date of perfused manometry is randomized to avoid bias due to examinations' order.
  Interventions: Device: Esophageal high resolution manometry associated or not with manometry with perfused Dentsleeve probe (as determined by randomization)

INTERVENTIONS:
Device: Esophageal high resolution manometry associated or not with manometry with perfused Dentsleeve probe (as determined by randomization) — Visit V0 (day 0 - 2 to 14 days):
  * Subject selection
  * Obtaining of written informed consent
  Visit V1 (day 0):
  * Fasting subject
  * Randomization to determine the examination order
  * Esophageal high resolution manometry (Sierra Scientific Instruments, California CA) associated or not with manometry with perfused Dentsleeve probe (as determined by randomisation): 3-hour recording (1 hour fasting, ingestion of a 600-kcal liquid meal in 10 minutes, 2 hours post prandial)
  Visit V2 (day 0 + 1 day): Phone contact
  Visit V3 (day 0 + 2 to 7 days):
  * Same as V1
  Visit V4 (V3 + 1 day): Phone contact and end of the study

SUMMARY:
Transient lower esophageal sphincter relaxations (tLESr) are the main mechanism of gastro-oesophageal reflux disease. They occur without any deglutition in patients but also in healthy volunteers. They are induced by meal.

The gold standard to detect tLESr is esophageal manometry using perfused Dentsleeve probe.

Esophageal high resolution manometry with solid state sensors was developed in the 90s. The examination is easier and more accurate than perfused manometry. The aim of this study is to validate in healthy volunteers the use of high resolution manometry (Sierra Scientific Instruments, California CA) to detect tLESr.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female between 18 and 60 years
2. Subject without typical or atypical symptoms of gastro-esophageal reflux disease (heartburn, regurgitation, epigastric pain, chest pain, chronic cough, pharyngeal pain)
3. Subject without any medication (except oral contraception)
4. Subject without previous digestive surgery history (except appendicectomy)
5. Capability to pass manometric probes through each nostril
6. Subject with health insurance
7. Written informed consent
8. No participation to another study at the same time

Exclusion Criteria:

1. Age under 18 years or upper 60
2. Pregnant woman or lactation
3. Incapability to give consent
4. No written informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to demonstrate that high resolution manometry allows the detection of meal-induced tLESr. All recordings will be analyzed at the end of each examination and reviewed at the end of the enrolment.

SECONDARY OUTCOMES:
To compare the number of tLESr detected by high resolution manometry and those detected by manometry with perfused dentsleeve probe.
To define the characteristics (duration, relaxation amplitude) of high resolution manometry-detected tLESr.

CONTACTS AND LOCATIONS:
Overall Officials: ROMAN Sabine, MD, Principal Investigator — Hospices Civils de Lyon; MION François, MD, Principal Investigator — Hospices Civils de Lyon; BRULEY DES VARANNES Stanislas, MD, Principal Investigator — CHRU NANTES; ZERBIB Frank, MD, Principal Investigator — CHRU BORDEAUX
Locations (3):
- France (3):
  - Hôpital St André, CHU BORDEAUX, Bordeaux
  - Hôpital Edouard Herriot - Hospices Civils de Lyon, Lyon
  - Hôpital Hôtel Dieu, CHU NANTES, Nantes